CLINICAL TRIAL: NCT05579652
Title: The Change in Tension of the Abdominal Wall Tension in Open Abdomens
Brief Title: Change in Fascial Tension in Open Abdomens
Status: Completed | Type: Observational
Sponsor: Benjamin T. Miller (Other)
Responsible Party: Sponsor-Investigator, Benjamin T. Miller, Assistant Professor, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: 22-845
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Abdominal Wall Defect; Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with open abdomen: All non-pregnant adults with an open abdomen who are consentable or who have a legally authorized representative will have the tension on each side of their abdominal wall measured using a tensiometer at each abdominal exploration
  Interventions: Diagnostic Test: Abdominal tension measurement

INTERVENTIONS:
Diagnostic Test: Abdominal tension measurement — A tensiometer scale will be used to measure the tension needed to pull each side of the abdominal wall to midline

SUMMARY:
The goal of this observational study is to quantitatively measure the change in tension of the abdominal wall over time in subjects with open abdomens using a tensiometer.

DETAILED DESCRIPTION:
For subjects undergoing damage control and decompressive laparotomy, surgeons frequently elect to keep the abdomen open in anticipation of multiple re-explorations or to prevent and/or treat abdominal compartment syndrome. The eventual goal is to definitively close the abdomen, including the fascia, when medically and surgically safe. The natural tendency with prolonged open abdomen is lateralization of the fascia, making closure of the fascia progressively more difficult as time passes. Though this is subjectively observed in the operating room as increased tension during fascial closure, there is no quantitative data describing how duration of open abdomen affects tension on the abdominal wall. This information has potential implications on the likelihood of successful primary closure, risk of dehiscence, and long term hernia development. This study aims to quantitatively measure the changes in tension of the abdominal wall over time in subjects with an open abdomen. A tensiometer will be used to measure the tension needed to approximate each side of the abdominal fascia to midline with each re-exploration until definitive abdominal wall closure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an open abdomen and plan for abdominal re-exploration

Exclusion Criteria:

* patients under the age of 18 years
* pregnant patients
* patients who have no available Legally Authorized Representative to provide consent.
* patients with a current hernia
* patients with a prior component separation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will identify patients with an open abdomen following laparotomy with plans to return to the operating room for re-exploration. Previous laparotomy, presence of a stoma, and presence of a previous hernia repair without component separation will not exclude patients from this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Change in tension over time | 1.5 years
  The progressive change in abdominal wall tension will be analyzed

SECONDARY OUTCOMES:
Subject factors affecting abdominal wall tension over time | 1.5 years
  Investigators will evaluate the relationship of BMI and age to the change in tension over time
Operative factors affecting abdominal wall tension over time | 1.5 years
  Investigators will evaluate the relationship of incision width and length, time in days that the abdomen was open, number of reoperations, and abdominal wall tension change over time.
Medical care factors affecting abdominal wall tension over time | 1.5 years
  Investigators will evaluate the relationship of volume and type of intravenous fluid administered, blood transfusion, diuresis, and vasopressor use and the change in abdominal wall tension over time.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Miller, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No